CLINICAL TRIAL: NCT01677299
Title: A Randomized, Crossover Study Assessing the Effects of pH 6.5 Enteric Coating of Metformin HCl Tablets on Pharmacokinetics and Changes in Circulating Glucose and Gastrointestinal Hormone Concentrations in Subjects With Type 2 Diabetes Mellitus
Brief Title: Assessing the PK and Effect on Glucose and GI Hormone Concentrations of Metformin Delayed-Release in Subjects With T2DM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elcelyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LCPOC10
Record Dates: First submitted 2012-08-23; First posted 2012-09-03 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1000 mg EFB0026 (metformin immediate-release) (Active Comparator): BID
  Interventions: Drug: EFB0026 (metformin immediate-release)
- 1000 mg EFB0027 (metformin delayed-release) (Experimental): BID
  Interventions: Drug: EFB0027 (metformin delayed release)
- 500 mg EFB0027 (metformin delayed-release) (Experimental): BID
  Interventions: Drug: EFB0027 (metformin delayed release)
- 500 mg EFB0026 + 1000 mg EFB0027 (Experimental): BID
  Interventions: Drug: EFB0027 (metformin delayed release); Drug: EFB0026 (metformin immediate-release)

INTERVENTIONS:
Drug: EFB0027 (metformin delayed release) — Comparison of enteric-coating to assess effect on PK
  Other Names: Met DR
  Arms: 1000 mg EFB0027 (metformin delayed-release); 500 mg EFB0026 + 1000 mg EFB0027; 500 mg EFB0027 (metformin delayed-release)
Drug: EFB0026 (metformin immediate-release) — Active comparator
  Other Names: Met IR; metformin; Glucophage
  Arms: 1000 mg EFB0026 (metformin immediate-release); 500 mg EFB0026 + 1000 mg EFB0027

SUMMARY:
This study will evaluate how EFB0027 and EFB0026 behave in subjects with type 2 diabetes mellitus.

In addition, this study will compare the effects of EFB0027 and EFB0026 on circulating concentrations of glucose and gastrointestinal hormones in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Is 19 to 70 (inclusive) years old at Visit 1 (Screening).
2. Is diagnosed with Type 2 Diabetes Mellitus with

   * HbA1c between 6.0 to 9.5% (inclusive) for subjects managing their diabetes with:

     i. Diet and exercise alone, or ii. A stable regimen (minimum of 2 months at Visit 1) of metformin alone, or iii. A stable regimen (minimum of 2 months at Visit 1) of DPP-4 inhibitor alone, OR
   * HbA1c between 6.0 to 8.5% (inclusive) for subjects managing their diabetes with a stable (minimum of 2 months at Visit 1) combination regimen of metformin and DPP-4 inhibitors.
3. Has serum creatinine below the upper limit of normal at Visit 1 and an estimated creatinine clearance above 80 using the Crockroft and Gault equation (CrCl = [(140 - age) x body weight in kg] / (serum creatinine x 72) x (0.85 for females) [ref. 3].
4. Has a body mass index (BMI) of 25.0 to 40.0 kg/m^2 (inclusive) at Screening.
5. Is male, or is female and meets all of the following criteria:

   * Not breastfeeding
   * Negative pregnancy test result (human chorionic gonadotropin, beta subunit) at Visit 1 (Screening) (not applicable to hysterectomized females)
   * Surgically sterile, postmenopausal, or if of childbearing potential, must practice and be willing to continue to practice appropriate birth control during the entire duration of the study
6. Has a physical examination with no clinically significant abnormalities as judged by the investigator.
7. Ability to understand and willingness to adhere to protocol requirements.
8. If on chronic thyroid pharmacologic therapy, the dose must be stable for at least 3 months prior to Visit 1 (Screening), and must have thyroid-stimulating hormone (TSH) test result in normal range at Visit 1 (Screening).

Exclusion Criteria:

1. Has a clinically significant medical condition that could potentially affect study participation and/or personal well-being, as judged by the investigator, including but not limited to the following conditions:

   * Hepatic disease
   * Renal disease
   * Gastrointestinal disease
   * Endocrine disorder except diabetes
   * Cardiovascular disease
   * Seizure disorder
   * Organ transplantation
   * Chronic infection
2. Has any chronic disease requiring medication that has been adjusted in the past 90 days (subjects may take acute intermittent over-the-counter medications such as Tylenol, if needed).
3. Has any drug treatment that affects gastric pH (prescription or over-the-counter), including any antacids or medications such as Rolaids or Pepcid within 2 days of Visit 1 (Screening).
4. Has had major surgery of any kind within 6 months of Visit 1 (Screening).
5. Has received a blood transfusion within 6 months of Visit 1 (Screening).
6. Has a history of >5 kg weight change within 3 months of Visit 1 (Screening).
7. Has clinical laboratory test (clinical chemistry, hematology, or urinalysis) abnormalities other than those expected in subjects with diabetes and judged by the investigator to be clinically significant at Visit 1 (Screening).
8. Has physical, psychological, or historical finding that, in the investigator's opinion, would make the subject unsuitable for the study.
9. Currently abuses drugs or alcohol or has a history of abuse that in the investigator's opinion would cause the individual to be noncompliant with study procedures.
10. Has donated blood within 2 months of Visit 1 (Screening) or is planning to donate blood during the study.
11. Has used insulin within 3 months of Visit 1 (Screening).
12. Has received GLP-1 receptor agonists and/or thiazolidinedione treatment within 6 months of Visit 1 (Screening).
13. Has known intolerance to metformin.
14. Has received any investigational drug within 1 month (or five half-lives of the investigational drug, whichever is greater) of Visit 1 (Screening).
15. Has known allergies or hypersensitivity to any component of study treatment.
16. Is employed by Elcelyx Therapeutics, Inc (that is an employee, temporary contract worker, or designee of the company).
17. Smokes more than 10 cigarettes per day, 2 cigars per day, or uses more than 1 can of smokeless tobacco per week.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Celerion, Inc., Tempe, Arizona
  - Celerion, Inc., Lincoln, Nebraska

REFERENCES:
- [Background] DeFronzo RA, Buse JB, Kim T, Burns C, Skare S, Baron A, Fineman M. Once-daily delayed-release metformin lowers plasma glucose and enhances fasting and postprandial GLP-1 and PYY: results from two randomised trials. Diabetologia. 2016 Aug;59(8):1645-54. doi: 10.1007/s00125-016-3992-6. Epub 2016 May 23. PMID 27216492

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: BCAD; Sequence 2: ABDC; Sequence 3: CDBA; Sequence 4: DACB: BID
  Treatment A = 1000 mg EFB0026 (Met IR) Treatment B = 1000 mg EFB0027 (Met DR) Treatment C = 500 mg EFB0027 (Met DR) Treatment D = 500 mg EFB0026 (Met IR) plus 1000 mg EFB0027 (Met DR)
Period: Overall Study
Arm/Group | Sequence 1: BCAD | Sequence 2: ABDC | Sequence 3: CDBA | Sequence 4: DACB
Started | 6 | 6 | 6 | 6
Completed | 6 | 3 | 5 | 5
Not Completed | 0 | 3 | 1 | 1
Not completed — Adverse Event | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sequence BCAD; Sequence ABDC; Sequence CDBA; Sequence DACB: A = 1000 mg EFB0026 BID B = 1000 mg EFB0027 BID C = 500 mg EFB0027 BID D = 500 mg EFB0026 BID plus 1000 mg EFB0027 BID
- Total: Total of all reporting groups
Arm/Group | Sequence BCAD | Sequence ABDC | Sequence CDBA | Sequence DACB | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (3.54) | 56.8 (7.22) | 49.7 (13.92) | 55.3 (7.79) | 51.3 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 4 | 12
  Male | 4 | 3 | 3 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 2
  White | 5 | 3 | 6 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 5 | 2 | 14
  Not Hispanic or Latino | 2 | 3 | 1 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 24
BMI [Mean (Standard Deviation); unit: kg/mˆ2] | 34.13 (5.455) | 30.67 (2.793) | 35.65 (2.935) | 32.87 (3.644) | 33.33 (4.05)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73 mˆ2] | 117.94 (22.065) | 114.65 (21.348) | 107.54 (16.644) | 93.43 (20.354) | 108.39 (21.161)
HbA1c [Mean (Standard Deviation); unit: %] | 7.62 (1.234) | 7.33 (0.965) | 8.07 (1.102) | 6.37 (.339) | 7.35 (1.108)
FPG [Mean (Standard Deviation); unit: mg/dL] | 182.5 (71.55) | 158 (42.96) | 179 (69.59) | 124.3 (15.03) | 161 (56.34)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (0-t) of Plasma Metformin
Description: Measures from the time of dosing (0 h) to the time of the last quantifiable concentration following dose administration. The dose of study medication was administered at t = -1 min relative to the start time of the standardized breakfast.
Time Frame: Time points at which data were collected to create the area under the curve (0-t) for plasma metformin were: t = -0.08, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, and 11 h relative to the start time of the standardized breakfast.
Population: Evaluable Population
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- 1000 mg EFB0026; 1000 mg EFB0027; 500 mg EFB0027; 500 mg EFB0026 + 1000 mg EFB0027: BID
Arm/Group | 1000 mg EFB0026 | 1000 mg EFB0027 | 500 mg EFB0027 | 500 mg EFB0026 + 1000 mg EFB0027
Number analyzed (Participants) | 19 | 19 | 19 | 19
ng*h/mL | 8672 (29.7) | 4774 (29.9) | 3842 (37.6) | 8075 (38.6)

2. Primary Outcome: Change in Fasting Plasma Glucose
Description: LS mean difference from Baseline (Day 1) to Day 5
Time Frame: Change from Baseline (Day 1) to Day 5
Population: Evaluable Population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- 1000 mg EFB0026: BID
  EFB0026: Active comparator
- 1000 mg EFB0027; 500 mg EFB0027: BID
  EFB0027: Comparison of enteric-coating to assess effect on PK
- 500 mg EFB0026 + 1000 mg EFB0027: BID
  EFB0027: Comparison of enteric-coating to assess effect on PK
  EFB0026: Active comparator
Arm/Group | 1000 mg EFB0026 | 1000 mg EFB0027 | 500 mg EFB0027 | 500 mg EFB0026 + 1000 mg EFB0027
Number analyzed (Participants) | 19 | 19 | 19 | 19
mg/dL | -22.5 (6.8) | -19.9 (5) | -16.4 (3.8) | -21.2 (4.7)
Statistical Analysis 1: Comparison: 1000 mg EFB0026; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Change in fasting plasma glucose from Baseline to Day 5 (end of treatment) for treatment A; LS mean diff (Day 5 - Baseline) = -22.5, 95% CI 2-sided [-37 to -8]
Statistical Analysis 2: Comparison: 1000 mg EFB0027; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Change in fasting plasma glucose from Baseline to Day 5 (end of treatment) for treatment B; LS mean diff (Day 5 - Baseline) = -20, 95% CI 2-sided [-30 to -9]
Statistical Analysis 3: Comparison: 500 mg EFB0027; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Change in fasting plasma glucose from Baseline to Day 5 (end of treatment) for treatment C; LS mean diff (Day 5 - Baseline) = -16, 95% CI 2-sided [-24 to -8]
Statistical Analysis 4: Comparison: 500 mg EFB0026 + 1000 mg EFB0027; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Change in fasting plasma glucose from Baseline to Day 5 (end of treatment) for treatment D; LS mean diff (Day 5 - Baseline) = -21, 95% CI 2-sided [-31 to -11]

3. Primary Outcome: Within Treatment Comparison Based on Ratios of AUCs of GLP-1
Time Frame: Ratio of Day 5 to Baseline
Population: Evaluable
Measure: Least Squares Mean (Standard Error); unit: none (values are ratios)
Arm/Group | 1000 mg EFB0026 | 1000 mg EFB0027 | 500 mg EFB0027 | 500 mg EFB0026 + 1000 mg EFB0027
Number analyzed (Participants) | 19 | 19 | 19 | 19
none (values are ratios) | 1.87 (0.18) | 1.62 (.11) | 1.69 (.15) | 1.88 (.19)
Statistical Analysis 1: Comparison: 1000 mg EFB0027; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Geometric LS mean ration = 1.6, 95% CI 2-sided [1.4 to 1.9]
Statistical Analysis 2: Comparison: 1000 mg EFB0026; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Geo LSmean ratio of (Day 5/Baseline) = 1.9, 95% CI 2-sided [1.5 to 2.3]
Statistical Analysis 3: Comparison: 500 mg EFB0027; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Geo LSmean ratio (Day 5/Baseline) = 1.7, 95% CI 2-sided [1.4 to 2.0]
Statistical Analysis 4: Comparison: 500 mg EFB0026 + 1000 mg EFB0027; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Geo LSmean ratio (Day 5/Baseline) = 1.9, 95% CI 2-sided [1.5 to 2.3]

4. Primary Outcome: Within Treatment Comparison Based on Ratios of AUCs of PYY
Time Frame: Ratio of Day 5 to Baseline
Population: Evaluable Population
Measure: Least Squares Mean (Standard Error); unit: none (values are ratios)
Arm/Group | 1000 mg EFB0026 | 1000 mg EFB0027 | 500 mg EFB0027 | 500 mg EFB0026 + 1000 mg EFB0027
Number analyzed (Participants) | 19 | 19 | 19 | 19
none (values are ratios) | 1.55 (.09) | 1.38 (.09) | 1.46 (.06) | 1.49 (.06)
Statistical Analysis 1: Comparison: 1000 mg EFB0026; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Geo LSmean ratio (Day 5/Baseline) = 1.5, 95% CI 2-sided [1.4 to 1.8]
Statistical Analysis 2: Comparison: 1000 mg EFB0027; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Geo LSmean ratio (Day 5/Baseline) = 1.4, 95% CI 2-sided [1.2 to 1.6]
Statistical Analysis 3: Comparison: 500 mg EFB0027; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Geo LSmean ratio (Day 5/Baseline) = 1.5, 95% CI 2-sided [1.3 to 1.6]
Statistical Analysis 4: Comparison: 500 mg EFB0026 + 1000 mg EFB0027; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Geo LSmean ratio (Day 5/Baseline) = 1.5, 95% CI 2-sided [1.4 to 1.6]

ADVERSE EVENTS:
Description: Population Intent to treat (ITT)
Groups:
- 1000 mg EFB0026 BID: A: Metformin immediate release BID
- 1000 mg EFB0027 BID: B: Metformin delayed release BID
- 500 mg EFB0027 BID: C: Metformin delayed release BID
- 500 mg EFB0026 BID Plus 1000 mg EFB0027 BID: D: Metformin immediate plus Metformin delayed release
Arm/Group | 1000 mg EFB0026 BID | 1000 mg EFB0027 BID | 500 mg EFB0027 BID | 500 mg EFB0026 BID Plus 1000 mg EFB0027 BID
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/20 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 6/22 | 5/20 | 4/20 | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1000 mg EFB0026 BID (N=22) | 1000 mg EFB0027 BID (N=20) | 500 mg EFB0027 BID (N=20) | 500 mg EFB0026 BID Plus 1000 mg EFB0027 BID (N=21)
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 — 3 periods completed: C,D,B. During washout period, the subject experienced severe cramping and throbbing pain on his right side and was hospitalized. The investigator assessed this event as not related to study medication.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1000 mg EFB0026 BID (N=22) | 1000 mg EFB0027 BID (N=20) | 500 mg EFB0027 BID (N=20) | 500 mg EFB0026 BID Plus 1000 mg EFB0027 BID (N=21)
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 3
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Gastrointestinal Stromal Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 0
Sinus Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study may be published by INSTITUTE, however the publication shall not disclose any SPONSOR Confidential Information, the INSTITUTE shall send the SPONSOR a copy of any such proposed publication 90 days prior to submission for publication, the INSTITUTE, on request of the SPONSOR, shall delete any SPONSOR Confidential Information in the proposed publication, and the INSTITUTE shall, on the SPONSOR's request, delay submission while the SPONSOR files applications for patents.